CLINICAL TRIAL: NCT02480894
Title: A Phase 1, Open-label, Drug-drug Interaction Study Between BMS-663068 and Maraviroc in Healthy Subjects
Brief Title: A Open-label, Drug-Drug Interaction With Maraviroc (DDI)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 206278; AI438-052 (Other: Bristol-Myers Squibb)
Record Dates: First submitted 2015-06-16; First posted 2015-06-25 (Estimated); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Infection, Human Immunodeficiency Virus
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome | interventions — fostemsavir; Maraviroc

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sequential Dosing (Experimental): Treatment A: BMS-663068 orally twice daily (BID) on Days 1 through 4 Treatment B: Maraviroc BID on Days 7 through 11 Treatment C: BMS-663068 BID plus maraviroc BID on Days 12 through 18
  Interventions: Drug: BMS-663068; Drug: Maraviroc

INTERVENTIONS:
Drug: BMS-663068 — BMS-663068
Drug: Maraviroc — Maraviroc

SUMMARY:
This is a Phase 1, open-label, single sequence, two-way interaction study in healthy male and female subjects. For the effect of maraviroc on the pharmacokinetics (PK) of BMS-626529 (the active moiety of BMS-663068), there is no formal hypothesis to be statistically tested. The purpose of this assessment is to estimate the effect of maraviroc on the PK of BMS-626529 when coadministered in healthy subjects. For the effect of BMS-663068 on the PK of maraviroc, the hypothesis to be statistically tested is that BMS-663068 will not have a clinically significant effect on the PK of maraviroc when coadministered in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female nonsmoking subjects ages 18 to 50 years, inclusive with a body mass index of 18.0 to 32.0 kg/m2, inclusive
* Women of childbearing potential must agree to follow instructions for methods of contraception for a total of 34 days post-treatment completion

Exclusion Criteria:

* Any condition possibly affecting drug absorption
* Pre-existing liver dysfunction
* Any significant acute or chronic medical illness
* Orthostatic intolerance
* Other protocol specified exclusion criteria could apply

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 112 (Actual)
Dates: Start 2015-07-07 (Actual); Primary Completion 2015-09-21 (Actual); Study Completion 2015-09-21 (Actual)

PRIMARY OUTCOMES:
BMS-626529 Pharmacokinetics: maximum observed plasma concentration (Cmax) | predose and up to 12 hours post dose on Days 4, 16, 17, and 18
  PK parameters for BMS-626529 in the absence or presence of multiple doses of maraviroc include:
  - Cmax
BMS-626529 Pharmacokinetics: area under the plasma concentration-time curve (AUC) in a single dosing interval AUC(TAU) | predose and up to 12 hours post dose on Days 4, 16, 17, and 18
  PK parameters for BMS-626529 in the absence or presence of multiple doses of maraviroc include:
  - AUC(TAU)
Maraviroc Pharmacokinetics: Cmax | predose and up to 12 hours post dose on Days 9, 10, 11, 16, 17, and 18
  PK parameters for maraviroc in the absence or presence of BMS-663068 include:
  - Cmax
Maraviroc Pharmacokinetics: AUC(TAU) | predose and up to 12 hours post dose on Days 9, 10, 11, 16, 17, and 18
  PK parameters for maraviroc in the absence or presence of BMS-663068 include:
  - AUC(TAU)

SECONDARY OUTCOMES:
Other PK Parameters for BMS-626529: Time of maximum observed plasma concentration (Tmax) | predose and up to 12 hours post dose on Days 4, 16, 17, and 18
  PK parameters for BMS-626529 include:
  - Tmax
Other PK Parameters for BMS-626529: plasma concentration observed at 12 hours post-dose (C12) | predose and up to 12 hours post dose on Days 4, 16, 17, and 18
  PK parameters for BMS-626529 include:
  - C12
Other PK Parameters for BMS-626529: trough observed plasma concentration (Ctrough) (predose) | predose and up to 12 hours post dose on Days 4, 16, 17, and 18
  PK parameters for BMS-626529 include:
  - Ctrough (predose)
Other PK Parameters for maraviroc: Tmax | predose and up to 12 hours post dose on Days 9, 10, 11, 16, 17, and 18
  PK Parameters for maraviroc include:
  -Tmax
Other PK Parameters for maraviroc: C12 | predose and up to 12 hours post dose on Days 9, 10, 11, 16, 17, and 18
  PK Parameters for maraviroc include:
  * C12
Other PK Parameters for maraviroc: Ctrough | predose and up to 12 hours post dose on Days 9, 10, 11, 16, 17, and 18
  PK Parameters for maraviroc include:
  - Ctrough
Clinical Safety as Measured by Adverse Events | Day 1 to Day 26
  Adverse event monitoring
Clinical Safety as Measured by Vital Signs | Day 1 to Day 26
  Vital sign measurement
Clinical Safety as Measured by Electrocardiograms (ECGs) | Day 1 to Day 26
  12-lead ECGs
Clinical Safety as Measured by Physical Examination | Day 1 to Day 26
  Physical examinations
Clinical Safety as Measured by Clinical Laboratory Evaluations | Day 1 to Day 26
  Clinical chemistry, hematology, urinalysis

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, San Antonio, Texas, United States

REFERENCES:
- [Derived] Wire MB, Magee M, Ackerman P, Llamoso C, Moore K. Evaluation of the pharmacokinetic drug-drug interaction between the antiretroviral agents fostemsavir and maraviroc: a single-sequence crossover study in healthy participants. HIV Res Clin Pract. 2021 Dec 9;23(1):1-8. Epub 2022 Mar 14. PMID 35285786